CLINICAL TRIAL: NCT01828892
Title: A Randomized Controlled Trial to Evaluate Fibrin Glue Application in the Treatment of Low-Output Enterocutaneous Fistulas
Brief Title: Glue Application in the Treatment of Low-Output Fistulas
Acronym: FG-treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Jianan Ren, Vice president of department of surgery, Jinling Hospital, Jinling Hospital, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20120819
Record Dates: First submitted 2013-04-01; First posted 2013-04-11 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-06

CONDITIONS: Low-output External Gastrointestinal Fistula
Keywords: Autologous platelet rich fibrin glue; Enterocutaneous fistulas; Single low output GI fistulas
MeSH Terms: conditions — Intestinal Fistula | interventions — Anti-Bacterial Agents; Ceftazidime; Cefotaxime; Meropenem; Nutrition Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PRFG treatment (Experimental): As described in our previous study, platelet-rich cryoprecipitate and thrombin were obtained from 300-400ml whole blood of each patient enrolled in the PRFG group and then frozen at -20°C for storage. Prior to application, frozen cryoprecipitate and thrombin stored were thawed in a 37°C water bath. Aminomethylbenzoic Acid (1ml: 1mg, Sigma-Aldrich, St Louis, MO) was added into the cryoprecipitate in the volume ratio of 1:10.
  Interventions: Procedure: Endoscopy exploration and glue application; Drug: Antibiotics (ceftazidime, cefotaxime, or meropenem, with or without vancomycin); Dietary Supplement: Nutrition support
- Control (Sham Comparator): Patients in this group only received standard of care when their fistula output < 200ml/24h.
  Interventions: Procedure: Endoscopy exploration; Drug: Antibiotics (ceftazidime, cefotaxime, or meropenem, with or without vancomycin); Dietary Supplement: Nutrition support
- Commercial FG (Experimental): Commercial FG (Zhejiang Puji Porcine fibrin sealant) was applied to close fistulas.
  Interventions: Procedure: Endoscopy exploration and glue application; Drug: Antibiotics (ceftazidime, cefotaxime, or meropenem, with or without vancomycin); Dietary Supplement: Nutrition support

INTERVENTIONS:
Procedure: Endoscopy exploration and glue application — A forward-viewing fistula-fiberscope (EndoView, Outai Medical Equipment, Shanghai, China), with 15cm length and 5mm width of fiber optical wire, was inserted into the fistula tract to accomplish endoscopic visualization. Briefly, the fistula-fiberscope assisted procedure was carried out percutaneously, allowing the exposure of internal hole and the whole tracts, followed by insertion of this catheter with distal mixing device.
  Arms: Commercial FG; PRFG treatment
Procedure: Endoscopy exploration — A forward-viewing fistula-fiberscope (EndoView, Outai Medical Equipment, Shanghai, China), with 15cm length and 5mm width of fiber optical wire, was inserted into the fistula tract to accomplish endoscopic visualization.
  Arms: Control
Drug: Antibiotics (ceftazidime, cefotaxime, or meropenem, with or without vancomycin) — Antibacterial therapy in patients with signs of systemic sepsis or local inflammation with pain
  Other Names: ceftazidime, cefotaxime, or meropenem, with or without vancomycin
Dietary Supplement: Nutrition support — Nutritional replacement and bowel rest via enteral or parenteral nutrition

SUMMARY:
Adjuvant use of fibrin glue (FG) in the fistula tract has been shown to promote closure of low-output enterocutaneous fistulas (ECFs). The primary objectives of this study are to compare the clinical efficacy, safety of autologous platelet-rich fibrin glue (PRFG), commercial fibrin glue, and control therapy in the management of patients with low-output volume ECFs.

DETAILED DESCRIPTION:
* This is a prospective, randomized, multi-centered study clinical, safety and economic outcome of ECFs patients.
* Subjects are randomized to one of 3 groups:

  * Group 1: Autologous PRFG-treatment [PRFG + Standard of care (SOC)]
  * Group 2: Commercial FG-treatment [FG + Standard of care (SOC)]
  * Group 3: Control (SOC only)
* Study will include three phases:

  * Phase 1: Screening, consent and enrollment
  * Phase 2: Patients will receive either PRFG, commercial FG, or SOC only for 14 days
  * Phase 3: Follow up: for patients with closed fistula within 14 days, we will follow up them for 6 months. For patients whose fistulas were still open will be treated with other therapeutic option and follow up for 6 months after closure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a single tubular ECF
* Low output volume (<200 ml/24h)
* Tract length >2cm
* Tract diameter < 1cm

Exclusion Criteria:

* Cancer-infiltrated fistula
* Abscess
* Foreign bodies
* Distal bowel obstruction
* Inflammatory Bowel Disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-03; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Closure rates up to 14 days | 14 days
  The fraction of patients with complete closure of fistula during 14 days

SECONDARY OUTCOMES:
Number of adverse events | Participants will be followed for at least 180 days
  Incidence of adverse events and severe adverse events up to 180 days (defined as an event that was fatal or life-threatening, led to additional hospitalization or disability, or required an intervention to prevent one of these outcomes)

OTHER OUTCOMES:
Economic outcome | From fistula onset to the end of treatment, which is at least 180 days
  Hospital cost upon enrollment, Hospital cost during entire hospital stay, Cost between fistula onset and final outcome

CONTACTS AND LOCATIONS:
Overall Officials: Jianan Ren, MD, Principal Investigator — Jinling Hospital, China
Locations (1):
- Jinling Hospital, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Wu X, Ren J, Wang G, Wang J, Wang F, Fan Y, Li Y, Han G, Zhou Y, Song X, Quan B, Yao M, Li J. Evaluating the use of fibrin glue for sealing low-output enterocutaneous fistulas: study protocol for a randomized controlled trial. Trials. 2015 Oct 7;16:445. doi: 10.1186/s13063-015-0966-9. PMID 26445823